CLINICAL TRIAL: NCT00243139
Title: A Randomized Controlled Trial of a Mandibular Advancement Device for Obstructive Sleep Apnea
Brief Title: Mandibular Advancement Device for Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nykøbing Falster County Hospital (Other)
Collaborators: University of Copenhagen (Other); Center of Expertise, Oringe Psychiatric Hospital,Vordingborg, Denmark (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNB01
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Sleep Apnea Syndromes; Sleep Apnea; Obstructive Sleep Apnea
Keywords: Oral appliances; Obstructive sleep apnea; Epworth Sleepiness Scale; SF-36
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Occlusal Splints

INTERVENTIONS:
Device: Mandibular advancement device (activator)

SUMMARY:
The purpose of this study was to determine how effective a custom-made standard dental splint (activator) advancing the lower jaw forward is in treatment of obstructive sleep apnea, and further to find factors for identification of those patients likely to benefit from this treatment.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is far the most common sleep disordered breathing, affecting 2-4% of the adult population. The repetitive obstructions are located in the pharyngeal airway, leading to sleep fragmentation and resulting in excessive daytime sleepiness with consequences for ability to work, road safety and quality of life. Furthermore, OSA is an independant riskfactor for cardiovascular disease. The treatment of choice today is continuous positive airway pressure (CPAP) but a main problem with CPAP is an unsatisfactory compliance. An alternative conservative more user-friendly treatment could be oral appliances, intending to increase the pharyngeal airway directly by tongue retaining devices or indirectly by mandibular advancing devices. Though several randomized studies on oral appliances have come recent years, all giving some evidence for effect on OSA, they all had some shortcomings, such as using crossover design, small sample sizes, under-reporting of methods and data and lack of blinding.

In this study of a mandibular advancement device was used a parallel group design with an inactive device and no intervention as controls. Beside the effect on sleep, daytime sleepiness and quality of life, the study aimed to find objective factors to be used as predictors of the outcome.

ELIGIBILITY:
Inclusion Criteria:

* AHI > 5 on polysomnography
* sufficient set of teeth to hold a splint
* written informed consent

Exclusion Criteria:

* sleep apnea with severe cardiovascular disease
* other severe somatic or psychiatric disease
* periodontal disease
* significant occlusal dysfunction
* pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 1999-07; Study Completion 2004-02

PRIMARY OUTCOMES:
Change in sleep parameters, especially apnea-hypopnea index (AHI).

SECONDARY OUTCOMES:
Change in daytime sleepiness, assessed by Epworth Sleepiness Scale.
Change in quality of life, assessed by SF-36.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Petri, MD, Principal Investigator — Nykoebing Falster County Hospital
Locations (1):
- Nykoebing Falster County Hospital, Nykoebing Falster, Storstrøms County, Denmark